CLINICAL TRIAL: NCT06763315
Title: The Efficacy, Safety, and Long-Term Prognosis of Low-Dose Selumetinib in the Treatment of Neurofibromatosis Type 1 Associated Plexiform Neurofibromas in Chinese Children: a Multicenter Randomized Controlled Trial
Brief Title: Low-dose Selumetinib for the Treatment of Plexiform Neurofibromas in Chinese Children
Acronym: LS-NF1PNs
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, Principal Investigator, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEL20241219
Record Dates: First submitted 2024-12-25; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Plexiform Neurofibromas (PN)
Keywords: Neurofibromatosis type 1; Plexiform neurofibromas; Selumetinib; Low-dose
MeSH Terms: conditions — Neurofibroma, Plexiform; Neurofibromatosis 1 | interventions — AZD 6244

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Regular dose of selumetinib (Active Comparator): The total daily dose is 25 mg/m², twice a day, once every 12 hours, and the treatment is continued and followed up for 24 cycles (28 days as one cycle).
  Interventions: Drug: Selumetinib
- Low dose of selumetinib (Experimental): The total daily dose is 20 mg/m², twice a day, once every 12 hours, and the treatment is continued and followed up for 24 cycles (28 days as one cycle).
  Interventions: Drug: Selumetinib

INTERVENTIONS:
Drug: Selumetinib — Use of the internationally recommended standard dose and low dose of the same drug
  Other Names: AZD6244; Koselugo

SUMMARY:
The goal of this study is to compare the efficacy and safety of low-dose and internationally recommended standard dose of selumetinib in the treatment of plexiform neurofibromas in Chinese children.

DETAILED DESCRIPTION:
Neurofibromatosis type 1 (NF1) is an autosomal dominant genetic disorder that affects multiple organ systems, with an estimated prevalence of approximately 1/3000. Around 50% of NF1 develop plexiform neurofibromas (PN), which can exhibit invasive growth, leading to compression of surrounding tissues. PN can progress rapidly within a short period, resulting in severe deformities and functional impairments that significantly impact the patient's quality of life.

In 2020, selumetinib was approved in the United States for the treatment of symptomatic PN patients aged ≥2 years who were ineligible for surgery, bringing new breakthroughs to this large patient population in China. In recent years, clinical trials have been conducted in many countries and regions to evaluate the efficacy and safety of selumetinib in the treatment of PN. Studies have demonstrated that after one year of treatment, 70% of patients achieved confirmed partial lesion reduction, accompanied by significant improvements in pain symptoms and quality of life. Furthermore, the safety was favorable, with 97.7% of adverse reactions classified as Grade I or II. In China, a single-arm clinical trial involving 16 children also showed that all patients had controlled lesions, of which 63% of children had confirmed partial relief. However, the current dosage for children in China refers to the recommended value of Phase I clinical trials (25 mg/m²) in the United States. There remains a lack of pharmacokinetic and pharmacodynamic data specific to the Chinese population. Since racial differences can influence drug metabolism, the current dosage may exceed the tolerance level for some Chinese children, potentially increasing the risk of serious adverse reactions. Clinically, families frequently report a high incidence of adverse effects such as paronychia, abdominal pain, and rash.

Therefore, conducting a dose optimization study based on the Chinese population and exploring the efficacy and safety of low-dose selumetinib in the treatment of PN in Chinese children is of great significance. These efforts will guide clinical practice, reduce adverse reactions, and enhance treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male and females;
* Between 3 and 18 years of age;
* Diagnosis of NF1 as determined by meeting at least 2 of the following 7 criteria: (1) six or more cafe-au-lait macules (greater than or equal to 0.5cm in prepubertal subjects or greater than or equal to1.5 cm in post pubertal subjects); (2) two or more neurofibromas (any type); (3) freckling in axilla or groin; (4) optic glioma; (5) two or more Lisch nodules; (6) a distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex); (7) a first-degree relative with NF1;
* Diagnosis of PN as determined by biopsy and pathological diagnosis;
* Complete resection of PN is not feasible without significant morbidity risk;
* Normal liver, kidney, and heart function;
* Previous treatment, last dose time: colony stimulating factor≥1 week, radiotherapy≥6 weeks, other study drugs>30 days;
* Able to undergo MRI evaluation;
* Consent of parents (or the person with parental authority in families): signed and dated written informed consent.

Exclusion Criteria:

* Patients with contraindications to selumetinib administration (e.g., allergy to selumetinib);
* Unable to swallow the entire selumetinib capsule;
* Ongoing hormone, immunotherapy, or chemotherapy for PN;
* Previously received multiple myelosuppressive chemotherapy regimens;
* Suffering from other severe and/or uncontrolled systemic diseases not related to NF1 (e.g., uncontrolled diabetes, hypertension, severe malnutrition, chronic liver or kidney disease, active gastrointestinal ulcers, etc.);
* Presence of optic nerve glioma, malignant glioma, malignant peripheral nerve sheath tumor, or other cancers requiring chemotherapy or radiotherapy;
* Presence of severe local or systemic uncontrolled infections;
* Impaired gastrointestinal function or chronic gastrointestinal diseases that may significantly affect the absorption of selumetinib;
* Patients with inadequate liver function: total bilirubin higher than or equal to 1.5 × the upper limit of the normal (ULN) for age and alanine aminotransferase and aspartate aminotransferase higher than or equal to 2.5 × the ULN for age;
* Patients with inadequate renal function: 3-5 years of age maximum serum creatinine (mg/dL) of 0.8; 6-10 years of age maximum serum creatinine (mg/dL) of 1.0; 11-18 years of age maximum serum creatinine (mg/dL) of 1.2;
* Insufficient bone marrow function: absolute neutrophil count lower than 1×109/L;
* Patients with cardiac insufficiency: echocardiogram shows abnormal ejection fraction;
* HIV-infected patients or patients with known immunodeficiency;
* Patients with a history of treatment with selumetinib or other MEK inhibitors;
* Patients who are unable to participate in treatment or follow-up evaluation plans during the study;
* Patients who are unable to give informed consent.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
The change in tumor volume of plexiform neurofibromas | Once every 3 cycles for the first 12 cycles, once every 6 cycles for the next 12 cycles (each cycle is 28 days).
  Treatment response was measured by volumetric magnetic resonance imaging (MRI) analysis performed at the start of treatment and after 3, 6, 9, 12, 18, and 24 cycles of treatment and independently assessed by 2 radiologists. Changes in PN size were categorized as further growth (increase of ≥20%), no change (<20% increase and <20% decrease), partial involution (decrease of ≥20% and <75%), nearly complete involution (decrease of ≥75% and <100%), or complete involution (100%).

SECONDARY OUTCOMES:
Frequency of adverse events | Once per cycle in the first 3 cycles, once every 3 cycles in the 4th to 12th cycles, and once every 6 cycles in the last 12 cycles (each cycle is 28 days).
  Frequency of adverse events (e.g. gastrointestinal disorders, eye disorders, skin disorders, paronychia, abnormal left ventricular ejection fraction, abnormal myocardial marker, abnormal liver function etc.) collected regularly during follow-up by the investigators and reported by the parents. All adverse events were collected and graded according to Common Terminology Criteria for Adverse Events, version 4.0 (CTCAE v4.0). The causality of the adverse event was determined by the multidisciplinary staff and was classified as definitively not related, probably not related, possibly related, probably related, or definitively related. Any dose reductions, interruptions, or cessations enacted at the discretion of the investigators were recorded.
Quality of life (QOL) in patients and their families | Once every 3 cycles for the first 12 cycles, once every 6 cycles for the next 12 cycles (each cycle is 28 days).
  The Pediatric Quality of Life Inventory (PedsQLTM) 4.0 was used. This genetic core scale is a multidimensional child self-report and parent proxy report measure that assesses health-related quality of life (QOL) in children, adolescents, and young adults aged 2 to 25 years. The PedsQL contains 23 global core measures of QOL, including subscales assessing four domains (physical, emotional, social, and school functioning).
The change of pain intensity | Once every 3 cycles for the first 12 cycles, once every 6 cycles for the next 12 cycles (each cycle is 28 days).
  The Numerical Rating Scale-11 (NRS-11) was used. This scale is a self-report measure that assesses pain intensity on an 11-point numeric scale. It consists of a horizontal line with 0 on the right end, representing "no pain," and 10 on the left end, representing "the worst pain you can imagine." Children aged 8 to 18 years were asked to circle a number from 0 to 10 that best described their worst pain in the past week, including: 1) self-selected most important tumor pain, 2) physician-selected target tumor pain, 3) overall tumor pain, and 4) other types of pain.
The change of pain interference | Once every 3 cycles for the first 12 cycles, once every 6 cycles for the next 12 cycles (each cycle is 28 days).
  The Pain Interference Index (PII) is a six-item measure that assesses the extent to which pain has interfered with daily activities over the past week, including concentration, spending time with friends, leisure and physical activities, mood, and sleep. The scale was slightly adapted after translation into English, and a parallel parent version was developed and validated in parents of children with chronic pain. In this study, children aged 8 to 18 years completed the self-report PII, and parents of children aged 5 to 18 years completed the parent-report PII. The total PII score is the average of all six items.
The change of physical functioning (mobility and upper extremity) | Once every 3 cycles for the first 12 cycles, once every 6 cycles for the next 12 cycles (each cycle is 28 days).
  The Patient-Reported Outcome Measurement Information System (PROMIS®) Physical Function Mobility and Upper Extremity 8-item short forms were used. This short form is used to assess the ability of a person to perform a variety of physical functions over the past 7 days, ranging from motor movements (e.g., standing up from the floor) to activities including self-care skills and vigorous exercise. Children aged 8-18 years completed the Pediatric Self-Report Short Form, and parents of children aged 5-18 years completed the parallel Parent Report Form. These PROMIS Physical Functioning Short Forms demonstrated good psychometric properties, including good reliability and construct validity in adolescents with a variety of medical conditions.
The change of neurocognitive abilities-attention and memory | Once every 3 cycles for the first 12 cycles, once every 6 cycles for the next 12 cycles(each cycle is 28 days).
  The Continuous Performance Test (CPT) was used. It assesses the subject's attention, response control, and sustained attention ability by presenting continuous visual or auditory stimuli and requiring the subject to respond according to specific rules. The test content usually includes quickly identifying specific stimuli and responding while ignoring other distracting stimuli. Evaluation indicators include reaction time, accuracy of correct responses, frequency of impulsive responses, and the individual's ability to maintain attention during the task, helping to identify attention deficits or response control problems.
The change of neurocognitive abilities-language ability | Once every 3 cycles for the first 12 cycles, once every 6 cycles for the next 12 cycles (each cycle is 28 days).
  Peabody Picture Vocabulary Test (PPVT) was used. It is a standardized tool for assessing an individual's vocabulary comprehension ability. It presents a set of pictures and verbal words and asks the subject to choose the picture that best matches the meaning of the word. The test covers words of varying difficulty and assesses an individual's auditory comprehension of words. The main evaluation indicators include language comprehension level, vocabulary, and cognitive ability, which help detect language development, language disorders, and intelligence level.
The change of neurocognitive abilities-executive function | Once every 3 cycles for the first 12 cycles, once every 6 cycles for the next 12 cycles (each cycle is 28 days).
  The Stroop test was used. It assesses an individual's inhibitory control and selective attention. It consists of two tasks: one is to ask the subject to report the font color of a word while ignoring the meaning of the word (color word task), and the other is to simply report the font color (simple color task). The test evaluates an individual's cognitive inhibition ability in conflict situations by comparing the performance of these two tasks. The main evaluation indicators include reaction time, task accuracy, and conflict inhibition ability.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ji, MD, PhD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gross AM, Dombi E, Wolters PL, Baldwin A, Dufek A, Herrera K, Martin S, Derdak J, Heisey KS, Whitcomb PM, Steinberg SM, Venzon DJ, Fisher MJ, Kim A, Bornhorst M, Weiss BD, Blakeley JO, Smith MA, Widemann BC. Long-term safety and efficacy of selumetinib in children with neurofibromatosis type 1 on a phase 1/2 trial for inoperable plexiform neurofibromas. Neuro Oncol. 2023 Oct 3;25(10):1883-1894. doi: 10.1093/neuonc/noad086. PMID 37115514
- [Background] Kim H, Yoon HM, Kim EK, Ra YS, Kim HW, Yum MS, Kim MJ, Baek JS, Sung YS, Lee SM, Lim HS, Lee BJ, Lim HT, Kim D, Yoon J, Bae H, Hwang S, Choi YH, Kim KA, Choi IH, Lee SW, Park SJ, Lee BH. Safety and efficacy of selumetinib in pediatric and adult patients with neurofibromatosis type 1 and plexiform neurofibroma. Neuro Oncol. 2024 Dec 5;26(12):2352-2363. doi: 10.1093/neuonc/noae121. PMID 38975694
- [Background] Gross AM, Glassberg B, Wolters PL, Dombi E, Baldwin A, Fisher MJ, Kim A, Bornhorst M, Weiss BD, Blakeley JO, Whitcomb P, Paul SM, Steinberg SM, Venzon DJ, Martin S, Carbonell A, Heisey K, Therrien J, Kapustina O, Dufek A, Derdak J, Smith MA, Widemann BC. Selumetinib in children with neurofibromatosis type 1 and asymptomatic inoperable plexiform neurofibroma at risk for developing tumor-related morbidity. Neuro Oncol. 2022 Nov 2;24(11):1978-1988. doi: 10.1093/neuonc/noac109. PMID 35467749
- [Background] Yang X, Yoo HK, Amin S, Cheng WY, Sundaresan S, Zhang L, Duh MS. Clinical and humanistic burden among pediatric patients with neurofibromatosis type 1 and plexiform neurofibroma in the USA. Childs Nerv Syst. 2022 Aug;38(8):1513-1522. doi: 10.1007/s00381-022-05513-8. Epub 2022 May 17. PMID 35579709
- [Background] Gross AM, Wolters PL, Dombi E, Baldwin A, Whitcomb P, Fisher MJ, Weiss B, Kim A, Bornhorst M, Shah AC, Martin S, Roderick MC, Pichard DC, Carbonell A, Paul SM, Therrien J, Kapustina O, Heisey K, Clapp DW, Zhang C, Peer CJ, Figg WD, Smith M, Glod J, Blakeley JO, Steinberg SM, Venzon DJ, Doyle LA, Widemann BC. Selumetinib in Children with Inoperable Plexiform Neurofibromas. N Engl J Med. 2020 Apr 9;382(15):1430-1442. doi: 10.1056/NEJMoa1912735. Epub 2020 Mar 18. PMID 32187457
- [Background] Dombi E, Baldwin A, Marcus LJ, Fisher MJ, Weiss B, Kim A, Whitcomb P, Martin S, Aschbacher-Smith LE, Rizvi TA, Wu J, Ershler R, Wolters P, Therrien J, Glod J, Belasco JB, Schorry E, Brofferio A, Starosta AJ, Gillespie A, Doyle AL, Ratner N, Widemann BC. Activity of Selumetinib in Neurofibromatosis Type 1-Related Plexiform Neurofibromas. N Engl J Med. 2016 Dec 29;375(26):2550-2560. doi: 10.1056/NEJMoa1605943. PMID 28029918